CLINICAL TRIAL: NCT04782661
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Study to Assess the Safety, Tolerability and Pharmacokinetics of JNJ-70075200 in Healthy Participants
Brief Title: A Study of JNJ-70075200 in Healthy Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Program terminated prior to enrolling subjects
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: CR108971; 2020-004946-12 (EudraCT Number); 70075200SLE1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-02-16; First posted 2021-03-04 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1: Single Ascending Dose (SAD) (Experimental): Participants will receive an oral solution of JNJ-70075200 or placebo in single ascending doses on Day 1 in cohorts 1, 2, 3, 4, 5a and 6 under fasted condition. Participants in cohort 5a will additionally receive the same study intervention under fed condition (Cohort 5b) after a washout period of at least 7 days.
  Interventions: Drug: JNJ-70075200; Drug: Placebo
- Part 2: Multiple Ascending Dose (MAD) (Experimental): After assessment of safety, tolerability and pharmacokinetics data in Part 1, participants will receive an oral solution of JNJ-70075200 or placebo twice daily in Cohorts 1 to 6 for 14 days under fasted/fed condition.
  Interventions: Drug: JNJ-70075200; Drug: Placebo
- Part 3: Single-dose Oral Solid Formulation (Optional) (Experimental): Participants will receive oral dose of JNJ-70075200 on Day 1 in Cohort 1 under fasted condition. Part 3 will start after obtaining a formal regulatory/ethical approval.
  Interventions: Drug: JNJ-70075200

INTERVENTIONS:
Drug: JNJ-70075200 — JNJ-70075200 solution or solid formulations will be administered orally.
Drug: Placebo — Placebo solution will be administered orally.
  Arms: Part 1: Single Ascending Dose (SAD); Part 2: Multiple Ascending Dose (MAD)

SUMMARY:
The purpose of the study is to evaluate safety and tolerability of JNJ-70075200 compared with placebo after administration of single ascending doses of JNJ-70075200 as oral solution (Part 1); multiple ascending doses of JNJ-70075200, administered as oral solution over 14 consecutive days (Part 2); and the option of a single dose of JNJ-70075200 administered as an oral solid formulation (Part 3).

ELIGIBILITY:
Inclusion criteria:

* Participants be healthy on the basis of physical examination, medical history, vital signs, and 12-lead Electrocardiogram (ECG) performed at screening. Any abnormalities, must be considered not clinically significant
* Participants be healthy on the basis of clinical laboratory tests performed at screening and Day -1. If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study
* No history of pathogen driven cancers (carcinomas, sarcomas, gastric cancer, bladder cancer,Cholangiocarcinoma)
* Body weight of at least 50 kilograms (kg) and body mass index (BMI) within the range 18 and 30 kilograms per square meter (kg/m^2) (BMI = weight/height^2) (inclusive)
* All women must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) at screening

Exclusion criteria:

* Participants having a history of liver or renal insufficiency (estimated creatinine clearance [CL] below 60 milliliter per minute [mL/min]); significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Participants having a QT interval corrected according to Fridericia's formula (QTcF) greater than (>) 450 milliseconds (msec) for males, and >470 msec for females, has a complete left or right bundle branch block, or has a history or current evidence of additional risk factors for torsades de pointes (for example, heart failure, hypokalemia, family history of Long QT Syndrome) at screening and at Day -1
* Known allergies, hypersensitivity, or intolerance to JNJ-70075200 or its excipients
* Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (for example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Participants having a history of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-V) criteria within 12 months before screening or positive test result(s) for alcohol or drugs of abuse (including barbiturates, opiates, cocaine, cannabinoids, amphetamines and benzodiazepines) at screening or Day -2

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-05-09 (Estimated); Study Completion 2022-09-23 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Treatment Emergent Adverse Events (TEAEs) | Up to 1 year and 1 month
  An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Percentage of Participants with Serious Adverse Events (SAEs) | Up to 1 year and 1 month
  A SAE is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a suspected transmission of any infectious agent via a medicinal product; is medically important.
Number of Participants with Clinically Significant Changes in Vital Signs | Up to 1 year and 1 month
  Number of participants with clinically significant changes in vital signs will be assessed.
Number of Participants with Clinically Significant Changes in Physical Examination | Up to 1 year and 1 month
  Number of participants with clinically significant changes in physical examination will be assessed.
Number of Participants With Clinically Significant Laboratory Abnormalities | Up to 1 year and 1 month
  Number of participants with clinically significant laboratory abnormalities related to hematology and clinical chemistry will be reported.
Change From Baseline in QTc Interval | Baseline, up to 1 year and 1 month
  Change from baseline in QT interval corrected for heart rate (QTc interval) using Fridericia method will be measured by electrocardiogram (ECG).
Change from Baseline in Heart Rate (HR) | Baseline, up to 1 year and 1 month
  Change from baseline in HR will be measured by ECG.
Change from Baseline in QRS Interval | Baseline, up to 1 year and 1 month
  Change from baseline in QRS interval will be measured by ECG.
Change from Baseline in PR Interval | Baseline, up to 1 year and 1 month
  Change from baseline in PR interval will be measured by ECG.
Change From Baseline in QT Interval | Baseline, up to 1 year and 1 month
  Change from baseline in QT interval will be measured by ECG.

SECONDARY OUTCOMES:
Part 1, 2 and 3: Plasma Concentration of JNJ-70075200 Over Time | Part 1 and Part 3: Predose, up to 72 hours postdose (up to Day 4), Part 2: Predose, up to 24 hours postdose (up to Day 15)
  Plasma samples will be analyzed to determine concentrations of JNJ-70075200 using a validated, specific, and sensitive liquid chromatography mass spectrometry/mass spectrometry (LC-MS/MS).
Part 1 and 3: Plasma Concentration of JNJ-70075200 Over Time (Food Effect) | Predose, up to 72 hours postdose (up to Day 4)
  Plasma samples will be analyzed to determine concentrations of JNJ-70075200 using a validated, specific, and sensitive LC-MS/MS.
Part 1 and 3: Percentage of Participants with TEAEs (Food Effect) | Up to 1 year and 1 month
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Part 1 and 3: Percentage of Participants with SAEs (Food Effect) | Up to 1 year and 1 month
  A SAE is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a suspected transmission of any infectious agent via a medicinal product; is medically important.
Part 1 and 3: Number of Participants with Clinically Significant Changes in Vital Signs (Food Effect) | Up to 1 year and 1 month
  Number of participants with clinically significant changes in vital signs will be assessed.
Part 1 and 3: Number of Participants with Clinically Significant Changes in Physical Examination (Food Effect) | Up to 1 year and 1 month
  Number of participants with clinically significant changes in physical examination will be assessed.
Part 1 and 3: Number of Participants With Clinically Significant Laboratory Abnormalities (Food Effect) | Up to 1 year and 1 month
  Number of participants with clinically significant laboratory abnormalities related to hematology and clinical chemistry will be reported.
Part 1 and 3: Change From Baseline in QTc Interval (Food Effect) | Baseline, up to 1 year and 1 month
  Change from baseline in QTc interval using Fridericia method will be measured by ECG.
Part 1 and Part 3: Change from Baseline in HR (Food Effect) | Baseline, up to 1 year and 1 month
  Change from baseline in HR will be measured by ECG.
Part 1 and Part 3: Change from Baseline in QRS Interval (Food Effect) | Baseline, up to 1 year and 1 month
  Change from baseline in QRS interval will be measured by ECG.
Part 1 and Part 3: Change from Baseline in PR Interval (Food Effect) | Baseline, up to 1 year and 1 month
  Change from baseline in PR interval will be measured by ECG.
Part 1 and Part 3: Change From Baseline in QT Interval (Food Effect) | Baseline, up to 1 year and 1 month
  Change from baseline in QT interval will be measured by ECG.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trials, Study Director — Janssen Research & Development, LLC
Locations (1):
- PRA Health Sciences Onderzoekscentrum Groningen, locatie Martini, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency